CLINICAL TRIAL: NCT07316530
Title: Clinical Investigation Exploring a Newly Developed Ostomy Baseplate.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CP381
Record Dates: First submitted 2025-11-25; First posted 2026-01-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-10

CONDITIONS: Stoma Ileostomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational device (Experimental): 1 day treatment with investigational device
  Interventions: Device: CP381
- Comparator (Active Comparator): 1 day treatment with comparator
  Interventions: Device: CP381

INTERVENTIONS:
Device: CP381 — All subjects will test the investigational device and the comparator for 6 hours during two different test days, with at least 14 days between the test days.
  Before the application of the investigational device as well as comparator, the stoma will be measured by the test personal and the baseplate will be pre-cut too big, leaving an approximately 5 mm distance from the edge of the hole in the baseplate to the stoma. The baseplates will be unique to each subject.

SUMMARY:
Peristomal skin complications (PSCs) are the predominant complication for people living with a stoma, which affect their quality of life negatively.

Among the main reasons for developing PSCs are that the peristomal skin is exposed to stomal output either due to leakage of output under the baseplate and/or imperfect cutting of the hole in the baseplate, and incorrect application creating a gap between the hole in the baseplate and the stoma.

To seal this gap, Coloplast has developed a new ostomy baseplate and the aim of the investigation is to explore the investigational device 's ability to help protect the peristomal skin.

ELIGIBILITY:
Inclusion Criteria:

* Has given written informed consent
* Is at least 18 years old
* Has full legal capacity
* Has an ileostomy with consistent liquid faecal output (6-7 Bristol scale).
* Has used flat SenSura Mio 1-piece or 2-piece for at least 14 days before the inclusion.
* Has had the stoma for at least 90 days
* Has a stoma size less than 45mm in diameter
* Has experienced symptoms of peristomal skin complications such as itching, burning, or pain in the peristomal area within the last 14 days
* Has suitable peristomal skin area (assessed by investigator) to participate in investigation
* Is willing to refrain from analgesics within 24 hours before the test days
* Is willing to refrain from antihistamine within 96 hours before the test days
* Is willing to refrain from steroid treatment within 24 hours before the test days

Exclusion Criteria:

* Is currently receiving or have within the past 60 days received radio-and/or chemotherapy.
* low doses radio- and/or chemotherapy (assessed by Principal Investigator) is allowed for other indications than cancer.
* Is currently receiving or have within the past 30 days received topical steroid treatment in the peristomal skin area, e.g., lotion or spray.
* Is breastfeeding
* Is pregnant based on urine pregnancy test.
* Has known hypersensitivity towards any of the devices used in the investigation.
* Participates in other clinical investigations. Exception: Participation in other Coloplast sponsored clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2025-11-03 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Maximum itching | 6 hours
  Maximum itching score between hour 4-6 after application of the investigational device and the comparator (scale from 0-10)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Krarup Simonsen, Humlebæk, Denmark